CLINICAL TRIAL: NCT02246426
Title: TRuSST: Treatment of Social Cognition in Schizophrenia Trial
Brief Title: Treatment of Social Cognition in Schizophrenia Trial
Acronym: TRuSST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Minnesota (Other); VA Greater Los Angeles Healthcare System (U.S. Federal Agency); University of California, Los Angeles (Other); Rush University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSC-1004-14; R44MH091793 (NIH)
Record Dates: First submitted 2014-09-16; First posted 2014-09-22 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Treatment (Experimental): Computerized plasticity-based adaptive cognitive training requiring a total maximum of 40 treatment sessions, 3-5 times weekly, 45-60 minutes per session.
  Interventions: Other: Computerized plasticity-based adaptive cognitive training
- Active Comparator (Active Comparator): Commercially available computerized training requiring a total maximum of 40 treatment sessions, 3-5 times weekly, 45-60 minutes per session.
  Interventions: Other: Commercially available computerized training

INTERVENTIONS:
Other: Computerized plasticity-based adaptive cognitive training — Computerized plasticity-based adaptive cognitive training for a total maximum of 40 treatment sessions, 3-5 times weekly, 40-60 minutes per session.
  Other Names: SocialVille
  Arms: Experimental Treatment
Other: Commercially available computerized training — Commercially available computerized training for a total maximum of 40 treatment sessions, 3-5 times weekly, 40-60 minutes per session.
  Arms: Active Comparator

SUMMARY:
This study is a multi-site, prospective, parallel arm, double-blind, randomized, controlled clinical trial to assess the efficacy of an experimental software program targeting social cognitive abilities versus a computer-based software control. Both the study and the software being investigated meet the criteria of Non-Significant Risk.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of SocialVille, an online training program we have recently developed (with support of a Phase I SBIR award) to treat the social cognition deficits evident in schizophrenia (DSM-IV ICD-9 Code 295.90).

SocialVille is a computerized, browser-playable program suite, designed to target information processing in the core social cognition domains of deficit in schizophrenia. It can be used from any internet-connected computer; through a dedicated clinician portal, the treating clinician can register users to treatment, continuously track and monitor their performance, and coach users throughout training. The specific aims of the study are:

1. Specific Aim 1: Evaluate the efficacy of SocialVille as a social cognition treatment in individuals with schizophrenia. We will conduct a large-scale, multi-site, double-blind, randomized controlled clinical trial of the SocialVille medical device vs. an active computer games control, which approximates challenge, computer time and interaction with experimenter. This large trial will be conducted at four sites: University of Minnesota Medical School (site PI: Dr. Sophia Vinogradov), the Greater Los Angeles VA (Dr. Michael Green), Rush University (Dr. Christine Hooker), and University of California, Los Angeles (Drs. Joseph Ventura and Keith Nuechterlein). Study participants will complete 30 hours of training from home. At baseline, mid-way through training and immediately following training, we will employ a structured assessment battery with a co-primary SC performance measure and a co-primary functional performance measure, as well as secondary measures of SC, functional capacity, functional outcome, motivation, and quality of life.
2. Specific Aim 2: Identify specific populations of treatment responders and non-responders. We will examine predictors of SC gain based on baseline participant demographic, symptom level, computer use, SC, and functional measures, as well as on learning rate and plateau performance measures derived over the course of SocialVille use to determine if it is possible to identify specific populations that respond very well to SocialVille use, or those who are unlikely to respond to SocialVille use.
3. Specific Aim 3: Evaluate the effects of training on the relatively distinct low vs. high-level social cognition constructs. We will separately examine the effects of training on the independent SC factors of low level social cue detection and high-level inferential process, correlated with clinical symptoms and functional outcome, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between 18 and 65 years old, inclusive, at the time of study screening
2. Subjects must have a diagnosis of schizophrenia as defined by an interview.
3. Subjects must demonstrate adequate decisional capacity, in the judgment of the consenting study staff member, to make a choice about participating in this research study.
4. Subjects must have been clinically stable (non-acute) for 8 weeks prior to consent; in the judgment of the Site Principal Investigator.
5. Subjects must have been maintained on a stable treatment of antipsychotics and/or other concomitant psychotropic treatment for at least 6 weeks prior to consent.
6. Subjects must have learned English before the age of 12 to ensure valid neuropsychological results.
7. Subjects must have the visual, auditory, and motor capacity to use the computerized intervention in the judgment of the consenting study staff person.
8. Subjects must have no more than a moderately severe rating on hallucinations and unusual thought content.

Exclusion Criteria:

1. Subjects should not have had a psychiatric hospitalization in the 8 weeks prior to consent.
2. Subjects who appear to be intoxicated or under the influence of a controlled substance on any day of assessment must be rescheduled or discontinued based upon the discretion of the site staff evaluator.
3. Subjects should not have a history of mental retardation or pervasive developmental disorder; or other neurological disorder (e.g., Traumatic Brain Injury, epilepsy, Parkinson's Disease.)
4. Subjects should not have been treated within 3 years of the date of consent with a computer-based cognitive training program manufactured by Posit Science.
5. Subjects should not be participating in a concurrent clinical trial that, in the judgment of the Site Principal Investigator, could affect the outcome of this one.
6. Subjects must not show suicidal ideation or behaviors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2015-03; Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Spatial Cognition (Multiple scores are aggregated to arrive at a single composite score) | At 6 weeks and At 12 weeks
  The a priori co-primary social cognitive outcome measure will be a composite score comprised of the following standardized, validated set of assessments:
  * Penn Emotion Recognition Test (ER40) - A test for visual emotion perception; total percent correct.
  * Prosody Identification (PROID) - A test for prosody identification; total percent correct.
  * Penn Facial Memory Test (PFMT) -Immediate recall. A test for immediate recall of faces; total percent correct.
  * Penn Facial Memory Test (PFMT) - Delayed recall. A test for delayed recall of faces; total percent correct.
  * Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT) - managing emotions subscale (D); correct responses.
  * The Empathic Accuracy (EA) scale; average correlation.
Change in Performance on the UCSD Performance-based Skills Assessment (Co-Primary Composite Measure) | At 6 weeks and At 12 weeks
  The a priori co-primary functional measure will be the functional capacity measure of The UCSD Performance-based Skills Assessment (UPSA) - total correct. Higher scores indicate better performance. We have chosen the UPSA since it is a well-validated measure frequently used in cognitive and SC training studies; In addition, it measures functional capacity, which is expected to be affected by SC change. The UPSA is designed to assess skills in five areas (Household Chores, Communication, Finance, Transportation, and Planning Recreational Activities) that reflect general abilities that are important components of independent living. Test-retest reliability ranged from .63-.80 over follow-up periods up to 36 months in patients with schizophrenia. Among patients, the UPSA performance correlated significantly with severity of negative symptoms and of cognitive impairment but not with that of positive or depressive symptoms.

SECONDARY OUTCOMES:
Symptoms utilizing the Positive and Negative Syndrome Scale | At 6 weeks and At 12 weeks
  Between-group magnitude of change in symptomatology utilizing the Positive and Negative Syndrome Scale (PANSS) - total score, negative symptoms, positive symptoms. Higher scores are indicative of greater symptomatology. The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of patients with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Negative subscale consists of 7 items which assesses the negative symptoms with subscale score ranging from 7 to 49, where higher score indicates greater severity.
Psychosocial Functioning utilizing the Global Functioning Scale | At 6 weeks and At 12 weeks
  Between-group magnitude of change in psychosocial functioning utilizing the Global Functioning Scale (GFS) - role and social subscales. Lower scores indicate greater impairment in functional performance. The Global Functioning Scale (GFS) is a clinician-administered questionnaire which is used to assess general psychosocial functioning. It is a 10-point rating scale (1-10), where lower score indicates greater impairment.
Social Functioning utilizing the Social Functioning Scale | At 6 weeks and At 12 weeks
  Between-group magnitude of change in social functioning utilizing the Social Functioning Scale (SFS). The Social Functioning Scale was constructed specifically to tap areas of social functioning that are crucial to the community maintenance of individuals with schizophrenia. The 7 domains include: social engagement/withdrawal, interpersonal behavior, pro-social activities, recreation, independence-competence, independence-performance, and employment/occupation. The raw scores for each domain are converted to scaled scores, with a mean of 100 and a standard deviation of 15. Higher scores are indicative of greater social functioning.
Independent Functioning utilizing the Specific Levels of Function | At 6 weeks and At 12 weeks
  Between-group magnitude of change in independent functioning utilizing the Specific Levels of Function (SLOF) - total score, as well as interpersonal, acceptability, activities, and work skills scores. The Specific Levels of Function (SLOF) is a 43-item scale designed to assess in detail an individual's basic living skills and level of independent functioning. Total score range from 43 to 215, higher scores indicate better functioning.
Functional Capacity utilizing Virtual Reality Functional Capacity Assessment | At 6 weeks and At 12 weeks
  Between-group magnitude of change in functional capacity - the Virtual Reality Functional Capacity Assessment (VRFCAT) - total completion time. The Virtual Reality Functional Capacity Assessment measures four different functional abilities: checking for the availability of items to complete a recipe, taking a bus, shopping in a store, and managing currency. The total time ranges from 0 - 60000ms.
Quality of Life utilizing the Quality of Life Scale | At 6 weeks and At 12 weeks
  Between-group magnitude of change in quality of life utilizing the Abbreviated Quality of Life Scale - total score as well as subscales. The Quality of Life Scale (QLS) is a scale commonly used as a measure of functioning in schizophrenia. The Abbreviated QLS (aQLS) includes 7 items representing all four interdependent theoretical constructs of the original 21-item QLS. Behavioral anchors are presented for each item, scored on a 0 (severe impairment) to 6 (high functioning) scale. Higher scores are indicative of greater quality of life.
Motivational systems utilizing Behavioral Inhibition/Behavioral Activation Scale | At 6 weeks and At 12 weeks
  Between-group magnitude of change in motivational systems utilizing the Behavioral Inhibition/Behavioral Activation Scale (BIS-BAS) - BAS drive, fun seeking, reward, and BIS scores. The Behavioral Inhibition/Behavioral Activation Scale is a 24-item self-report questionnaire designed to assess the two general motivational systems that underlie behavior and affect, i.e. sensitivity to anticipated punishment or reward. Higher scores indicate greater sensitivity to punishment or reward.
Pleasure utilizing the Temporal Experience of Pleasure Scale | At 6 weeks and At 12 weeks
  Between-group magnitude of change in pleasure utilizing the Temporal Experience of Pleasure Scale (TEPS) - total scores. The Temporal Experience of Pleasure Scale is a measure specifically designed to capture the anticipatory (10 items) and consummatory (8 items) facets of pleasure. It is a 6-point Likert scale from 1 (very false for me) to 6 (very true for me). Higher scores indicate greater pleasure experience.
Social Perception utilizing The Awareness of Social Inference Test | At 6 weeks and At 12 weeks
  Between-group magnitude of change in social perception utilizing The Awareness of Social Inference Test (TASIT; Part 3) - total score. The Awareness of Social Inference Test Part 3 assesses the ability to differentiate between different kinds of counterfactual comments (lies and sarcasm). Scores range from 0-65 with lower scores indicating greater impairment in social functioning.
Emotion Perception utilizing the Morphed Faces Task | At 6 weeks and At 12 weeks
  Between-group magnitude of change in emotion perception utilizing the Morphed Faces Task - accuracy and reaction time. The Morphed Faces Task is a computerized emotion perception task, in which participants are presented with faces that are morphed between a neutral expression and an emotional expression (happy, disgusted, angry, or fearful).
Theory of Mind utilizing the Faux Pas Test | At 6 weeks and At 12 weeks
  Between-group magnitude of change in theory of mind utilizing the Faux Pas Test - total score. This test uses 5/10 faux pas stories and 5/10 control stories from the original Faux Pas Test. After each story is read, participants will be asked five questions for: detecting a faux pas, understanding the faux pas, understanding the mental state of the faux pas recipient, understanding the mental state of the person delivering the faux pas and understanding the details but without making inferences about the mental states of the characters in the story. The Faux Pas Test is a Theory of Mind (ToM) measure, which includes 20 short stories, incidents of faux pas (someone mistakenly saying something they shouldn't have). Lower scores indicate poor performance on the task.
Source Memory utilizing Source Memory Test | At 6 weeks and At 12 weeks
  Between-group magnitude of change in source memory utilizing the Source Memory Test - Hit and False Alarm Rates. The Source Memory Test is measure of memory for the source of self-generated, and experimenter-provided word items that shows strong associations to social cognition.
Hostility Bias utilizing Ambiguous Intentions Hostility Questionnaire | At 6 weeks and At 12 weeks
  Between-group magnitude of change in hostility bias utilizing the Ambiguous Intentions Hostility Questionnaire (AIHQ) - total score. The Ambiguous Intentions Hostility Questionnaire is a measure of attributional style, and specifically of hostile social-cognitive biases comprised of a variety of negative situations that differ in terms of intentionality. Higher scores indicate increased tendency to see other's action as hostile.

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Lee, PhD, Principal Investigator — Posit Science Corporation
Locations (4):
- United States (4):
  - Greater Los Angeles VA, Los Angeles, California
  - UCLA, Los Angeles, California
  - Rush University, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- [Derived] Roberts MT, Lloyd J, Valimaki M, Ho GW, Freemantle M, Bekefi AZ. Video games for people with schizophrenia. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD012844. doi: 10.1002/14651858.CD012844.pub2. PMID 33539561
- [Derived] Nahum M, Lee H, Fisher M, Green MF, Hooker CI, Ventura J, Jordan JT, Rose A, Kim SJ, Haut KM, Merzenich MM, Vinogradov S. Online Social Cognition Training in Schizophrenia: A Double-Blind, Randomized, Controlled Multi-Site Clinical Trial. Schizophr Bull. 2021 Jan 23;47(1):108-117. doi: 10.1093/schbul/sbaa085. PMID 32614046
- [Derived] Rose A, Vinogradov S, Fisher M, Green MF, Ventura J, Hooker C, Merzenich M, Nahum M. Randomized controlled trial of computer-based treatment of social cognition in schizophrenia: the TRuSST trial protocol. BMC Psychiatry. 2015 Jul 3;15:142. doi: 10.1186/s12888-015-0510-1. PMID 26138715